CLINICAL TRIAL: NCT02780115
Title: A Phase 2, Multicenter, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety, Efficacy, and Pharmacokinetics of the Fixed Combination of AGN-199201 and AGN-190584 in Patients With Presbyopia
Brief Title: A Safety, Efficacy and Pharmacokinetic Study of AGN-199201 and AGN-190584 in Patients With Presbyopia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 199201-010
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: Vehicle Control (Experimental): Vehicle dosed in both eyes administered once daily during office visits 1 through 5.
  Interventions: Drug: AGN-199201 Vehicle; Drug: AGN-190584 Vehicle
- Cohort 2: AGN-199201 Dose A and AGN-190584 Dose A (Experimental): Fixed combinations of AGN-199201 Dose A and AGN-190584 Dose A dosed in both eyes administered once daily during office visits 1 through 5.
  Interventions: Drug: AGN-199201 ophthalmic solution; Drug: AGN-190584 ophthalmic solution
- Cohort 3: AGN-199201 Dose B and AGN-190584 Dose B (Experimental): Fixed combinations of AGN-199201 Dose B and AGN-190584 Dose B dosed in both eyes administered once daily during office visits 1 through 5.
  Interventions: Drug: AGN-199201 ophthalmic solution; Drug: AGN-190584 ophthalmic solution
- Cohort 4: AGN-199201 Dose C and AGN-190584 Dose C (Experimental): Fixed combinations of AGN-199201 Dose C and AGN-190584 Dose C dosed in both eyes administered once daily during office visits 1 through 5.
  Interventions: Drug: AGN-199201 ophthalmic solution; Drug: AGN-190584 ophthalmic solution
- Cohort 5: Vehicle, AGN-199201 Dose C and AGN-190584 Dose C (Experimental): Dominant eye dosed with Vehicle. Fixed combinations of AGN-199201 Dose C and AGN-190584 Dose C dosed in nondominant eye. Treatment administered once daily during office visits 1 through 5.
  Interventions: Drug: AGN-199201 ophthalmic solution; Drug: AGN-190584 ophthalmic solution; Drug: AGN-199201 Vehicle; Drug: AGN-190584 Vehicle

INTERVENTIONS:
Drug: AGN-199201 ophthalmic solution — 1 drop of AGN-199201 ophthalmic solution Doses A, B, C in the eye.
  Arms: Cohort 2: AGN-199201 Dose A and AGN-190584 Dose A; Cohort 3: AGN-199201 Dose B and AGN-190584 Dose B; Cohort 4: AGN-199201 Dose C and AGN-190584 Dose C; Cohort 5: Vehicle, AGN-199201 Dose C and AGN-190584 Dose C
Drug: AGN-190584 ophthalmic solution — 1 drop of AGN-190584 ophthalmic solution Doses A, B, C in the eye.
  Arms: Cohort 2: AGN-199201 Dose A and AGN-190584 Dose A; Cohort 3: AGN-199201 Dose B and AGN-190584 Dose B; Cohort 4: AGN-199201 Dose C and AGN-190584 Dose C; Cohort 5: Vehicle, AGN-199201 Dose C and AGN-190584 Dose C
Drug: AGN-199201 Vehicle — Vehicle to AGN-199201
  Arms: Cohort 1: Vehicle Control; Cohort 5: Vehicle, AGN-199201 Dose C and AGN-190584 Dose C
Drug: AGN-190584 Vehicle — Vehicle to AGN-190584
  Arms: Cohort 1: Vehicle Control; Cohort 5: Vehicle, AGN-199201 Dose C and AGN-190584 Dose C

SUMMARY:
This is a safety, efficacy and pharmacokinetics study of the fixed combination of AGN-199201 and AGN-190584 in participants with presbyopia (inability to focus on items close-up).

ELIGIBILITY:
Inclusion Criteria:

* Normal vision at distance, either natural or post corneal laser refractive surgery, with presbyopia in each eye and complaints of poor near vision that impacts activities of daily living

Exclusion Criteria:

* Use of any topical ophthalmic medications, including artificial tears other than the study medications during the study
* Corneal abnormalities in either eye that interfere with visual acuity
* History of cataract surgery, phakic intraocular lens surgery, corneal inlay surgery or any intraocular surgery
* Diagnosis of glaucoma or ocular hypertension.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haixia Liu, Study Director — Allergan
Locations (25):
- United States (25):
  - Retina Institute of California Medical Group, Arcadia, California
  - Sall Research Medical Center, Artesia, California
  - WCCT Global, LLC, Cypress, California
  - Specialty Eye Care Medical Center, Glendale, California
  - Lugene Eye Institute, Glendale, California
  - The Eye Research Foundation, Newport Beach, California
  - Stanford Eye and Laser Center, Palo Alto, California
  - Wolstan and Golberg Eye Associates, Torrance, California
  - MedEye Associates, Miami, Florida
  - Central Florida Eye Institute, Ocala, Florida
  - Center for Sight, Sarasota, Florida
  - Clayton Eye Center, Morrow, Georgia
  - Silverstein Eye Centers, Louisville, Kentucky
  - The Eye Care Institute, Louisville, Kentucky
  - Specialized Eye Care, Baltimore, Maryland
  - James D. Branch, Winston-Salem, North Carolina
  - Devers Eye Institute, Portland, Oregon
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Total Eye Care, PA, Memphis, Tennessee
  - Cataract and Glaucoma Center, El Paso, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - R and R Eye Research, LLC, San Antonio, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Hoopes Durrie Rivera Research, LLC, Draper, Utah

REFERENCES:
- [Derived] Shirneshan E, Coon CD, Johnson N, Stokes J, Wells T, Lundy JJ, Andrae DA, Evans CJ, Campbell J. Development of the Near Vision Presbyopia Task-based Questionnaire for use in evaluating the impact of presbyopia. J Patient Rep Outcomes. 2021 Dec 2;5(1):125. doi: 10.1186/s41687-021-00378-y. PMID 34855038
- [Derived] Johnson N, Shirneshan E, Coon CD, Stokes J, Wells T, Lundy JJ, Andrae DA, Evans CJ, Campbell J. Development of the Presbyopia Impact and Coping Questionnaire. Ophthalmol Ther. 2021 Dec;10(4):1057-1075. doi: 10.1007/s40123-021-00391-w. Epub 2021 Oct 13. PMID 34643894

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization and treatment assignment were based on a randomization scheme prepared by Allergan Biostatistics prior to the start of the study.
Groups:
- Cohort 2: AGN-199201 Lower Dose and AGN-190584 Lower Dose: Fixed combinations of AGN-199201 Lower Dose and AGN-190584 Lower Dose dosed in both eyes administered once daily during office visits 1 through 5.
- Cohort 3: AGN-199201 Medium Dose and AGN-190584 Medium Dose: Fixed combinations of AGN-199201 Medium Dose and AGN-190584 Medium Dose dosed in both eyes administered once daily during office visits 1 through 5.
- Cohort 4: AGN-199201 Higher Dose and AGN-190584 Higher Dose: Fixed combinations of AGN-199201 Higher Dose and AGN-190584 Higher Dose dosed in both eyes administered once daily during office visits 1 through 5.
- Cohort 5: Vehicle, AGN-199201 Higher Dose and AGN-190584 Higher Dose: Dominant eye dosed with Vehicle. Fixed combinations of AGN-199201 Higher Dose and AGN-190584 Higher Dose dosed in nondominant eye. Treatment administered once daily during office visits 1 through 5.
Period: Overall Study
Arm/Group | Cohort 1: Vehicle Control | Cohort 2: AGN-199201 Lower Dose and AGN-190584 Lower Dose | Cohort 3: AGN-199201 Medium Dose and AGN-190584 Medium Dose | Cohort 4: AGN-199201 Higher Dose and AGN-190584 Higher Dose | Cohort 5: Vehicle, AGN-199201 Higher Dose and AGN-190584 Higher Dose
Started | 28 | 30 | 30 | 32 | 31
Completed | 28 | 29 | 29 | 31 | 30
Not Completed | 0 | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: All patients who received ≥ 1 administration of study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Vehicle Control | Cohort 2: AGN-199201 Lower Dose and AGN-190584 Lower Dose | Cohort 3: AGN-199201 Medium Dose and AGN-190584 Medium Dose | Cohort 4: AGN-199201 Higher Dose and AGN-190584 Higher Dose | Cohort 5: Vehicle, AGN-199201 Higher Dose and AGN-190584 Higher Dose | Total
Number analyzed (Participants) | 28 | 30 | 30 | 32 | 31 | 151
Age, Continuous [Median (Standard Deviation); unit: Years] | 48.3 (3.9) | 49.4 (2.7) | 47.9 (3.9) | 49.2 (3.8) | 48.1 (3.4) | 48.6 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 18 | 25 | 23 | 105
  Male | 9 | 10 | 12 | 7 | 8 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 11 | 9 | 14 | 53
  Not Hispanic or Latino | 19 | 20 | 19 | 23 | 17 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 0 | 2
  Asian | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 3 | 5 | 5 | 8 | 4 | 25
  White | 23 | 23 | 25 | 23 | 26 | 120
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Baseline UNVA severity [Count of Participants; unit: Participants] — Baseline UNVA measured visual acuity using Snellen Scores. Worse "severity" meant poorer visual acuity as measured by baseline UNVA (uncorrected near visual acuity). This graded measure was used to stratify participants into two groups: UNVA at baseline (≤ 20/80 and > 20/80).
  Participants
    ≤ 20/80 | 20 | 20 | 18 | 19 | 22 | 99
    > 20/80 | 8 | 10 | 12 | 13 | 9 | 52

OUTCOME MEASURES:

1. Primary Outcome: Weighted Average Change From Baseline in Uncorrected Near Visual Acuity (UNVA) Letters in the Nondominant Eye
Description: UNVA is assessed without corrective lenses in the non-dominant eye. UNVA is measured using an eye chart and is reported as the number of lines read correctly. The lower the number of lines read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of lines read correctly means that vision has improved.
Time Frame: Baseline, Day 28
Population: Modified Intent-to-Treat (mITT) population: all randomized patients who were randomized with a baseline and at least 1 post baseline assessment of mesopic, high contrast, UNVA.
Measure: Least Squares Mean (Standard Error); unit: letters correctly read
Arm/Group | Cohort 1: Vehicle Control | Cohort 2: AGN-199201 Lower Dose and AGN-190584 Lower Dose | Cohort 3: AGN-199201 Medium Dose and AGN-190584 Medium Dose | Cohort 4: AGN-199201 Higher Dose and AGN-190584 Higher Dose | Cohort 5: Vehicle, AGN-199201 Higher Dose and AGN-190584 Higher Dose
Number analyzed (Participants) | 28 | 30 | 30 | 32 | 31
letters correctly read | 3.00 (1.03) | 4.96 (1.00) | 7.77 (1.00) | 7.54 (0.97) | 7.81 (1.02)
Statistical Analysis 1: Comparison: Cohort 2: AGN-199201 Lower Dose and AGN-190584 Lower Dose; Test type: Superiority; p = 0.1663, ANCOVA; LS Mean Diff = 1.96, 95% CI 2-sided [-0.83 to 4.74]
Statistical Analysis 2: Comparison: Cohort 3: AGN-199201 Medium Dose and AGN-190584 Medium Dose; Test type: Superiority; p = 0.0009, ANCOVA; LS Mean Diff = 4.77, 95% CI 2-sided [1.98 to 7.56]
Statistical Analysis 3: Comparison: Cohort 4: AGN-199201 Higher Dose and AGN-190584 Higher Dose; Test type: Superiority; p = 0.0014, ANCOVA; LS Mean Diff = 4.54, 95% CI 2-sided [1.79 to 7.29]
Statistical Analysis 4: Comparison: Cohort 5: Vehicle, AGN-199201 Higher Dose and AGN-190584 Higher Dose; Test type: Superiority; p = 0.0008, ANCOVA; LS Mean Diff = 4.81, 95% CI 2-sided [2.03 to 7.58]

2. Secondary Outcome: Number of Participants Experiencing One or More Treatment Emergent Adverse Events (TEAEs)
Description: A Treatment Emergent Adverse Event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. An Adverse Drug Reaction was a harmful and unintended reaction that is incurred during routine administration or use of the drug, whose causal relationship with the drug cannot be excluded.
Time Frame: up to 65 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Vehicle Control | Cohort 2: AGN-199201 Lower Dose and AGN-190584 Lower Dose | Cohort 3: AGN-199201 Medium Dose and AGN-190584 Medium Dose | Cohort 4: AGN-199201 Higher Dose and AGN-190584 Higher Dose | Cohort 5: Vehicle, AGN-199201 Higher Dose and AGN-190584 Higher Dose
Number analyzed (Participants) | 28 | 30 | 30 | 32 | 31
Participants | 8 | 12 | 15 | 15 | 10

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for up to 65 days.
Description: Safety population: All patients who received ≥ 1 administration of study treatment
Arm/Group | Cohort 1: Vehicle Control | Cohort 2: AGN-199201 Lower Dose and AGN-190584 Lower Dose | Cohort 3: AGN-199201 Medium Dose and AGN-190584 Medium Dose | Cohort 4: AGN-199201 Higher Dose and AGN-190584 Higher Dose | Cohort 5: Vehicle, AGN-199201 Higher Dose and AGN-190584 Higher Dose
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30 | 0/30 | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30 | 0/30 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 7/28 | 8/30 | 10/30 | 11/32 | 7/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Vehicle Control (N=28) | Cohort 2: AGN-199201 Lower Dose and AGN-190584 Lower Dose (N=30) | Cohort 3: AGN-199201 Medium Dose and AGN-190584 Medium Dose (N=30) | Cohort 4: AGN-199201 Higher Dose and AGN-190584 Higher Dose (N=32) | Cohort 5: Vehicle, AGN-199201 Higher Dose and AGN-190584 Higher Dose (N=31)
Vision blurred (Eye disorders) | 0 | 2 | 3 | 3 | 2
Instillation site pruritus (General disorders) | 0 | 4 | 0 | 1 | 2
Instillation site foreign body sensation (General disorders) | 3 | 3 | 1 | 0 | 1
Instillation site pain (General disorders) | 3 | 4 | 1 | 3 | 1
Instillation site lacrimation (General disorders) | 3 | 3 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 5 | 1 | 1
Headache (Nervous system disorders) | 3 | 5 | 6 | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT02780115/SAP_000.pdf
  • Study Protocol (2016-08-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT02780115/Prot_001.pdf